CLINICAL TRIAL: NCT00461994
Title: The Role of Exercise and/or Diet in Weight Loss, and Weight Maintenance in Obese Preadolescent Children
Brief Title: The Role of Exercise and Diet in Weight Loss in Obese Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Collaborators: D-Cure, Israel (Industry); Soroka University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rmc003189CTil
Record Dates: First submitted 2007-04-17; First posted 2007-04-18 (Estimated); Last update posted 2007-04-18 (Estimated); Status verified 2007-04

CONDITIONS: Pediatric Obesity
Keywords: OBESITY; CHILDREN; METABOLIC PARAMETERS; DIET; EXERCISE
MeSH Terms: conditions — Pediatric Obesity; Obesity; Motor Activity | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: diet
Behavioral: exercise
Behavioral: diet and exercise

SUMMARY:
A 3-arms randomized prospective intervention study to determine the roles of exercise and/or diet on weight loss and weight maintenance in obese preadolescent children 6-11 year-old with BMI> 95th percentile for age and gender. Children were randomly allocated into three groups. The first group underwent an exercise program, the second one underwent both an exercise program and a diet program and the third underwent a diet program alone.

The total duration of the intervention is 12 weeks followed by a period of 9 months of follow-up. The effects of the different intervention on weight loss and weight maintenance,body composition, on hormonal components that regulate the caloric balance, on metabolic profile and cardiovascular risk factors and on psychological parameters were also determined.

DETAILED DESCRIPTION:
A 3-arms randomized prospective intervention study including 161 patients in order to determine the roles of exercise and/or diet on weight loss and weight maintenance in obese preadolescent children 6-11 year-old with BMI> 95th percentile for age and gender. The study recruited patients from 2 endocrine clinics.

Objectives:

1. The main aim was to determine the roles of exercise and/or diet on weight loss and weight maintenance in obese children.
2. Secondary goals were:

   1. To determine the effects of exercise and/or diet on body composition.
   2. To determine the effects of exercise and/or diet on leptin and ghrelin that play a role in the regulation of energy balance.
   3. To determine the effects of exercise and/or diet on metabolic profile, cardiovascular risk factors, and inflammatory markers as fasting glucose,insulin and lipid profile,homocysteine ,adiponectin levels,CRP,and IL-6.
   4. To determine the role of exercise and/or diet on psychological parameters of obese children.

Study Population

Inclusion Criteria

1. Obese preadolescent children 6-11 year-old with BMI> 95th percentile for age and gender.
2. A signed informed consent will be taken from patients and their parents.
3. Agreement to a follow-up of one year.

Exclusion Criteria

1. Cardiac problems (arrhythmia, Congestive heart disease)
2. Uncontrolled hypertension
3. Severe hepatic impairment (liver enzymes above 3 folds the upper normal values)
4. Renal failure
5. Genetic syndromes associated with obesity
6. Presence of untreated hypothyroidism
7. Participation in a clinical study during the last month methods Children fulfilling the inclusion and exclusion criteria were randomly allocated into one of three groups.

The first group underwent an exercise program, the second one underwent both an exercise program and a diet program and the third underwent a diet program alone.

On the first visit of the study, at the end of the intervention (12 weeks) and at the end of the follow-up period (1 year) the following had been checked:

Weight, Height, Body impedance, Waist and hip circumferences, Skin-folds, Blood pressure, Basal Metabolic Rate (evaluated by a metabolic monitor), and blood samples for: Blood count, Liver function, Renal function, Fasting Lipid, glucose and insulin,CRP, IL-6, TSH, free T4, Homocysteine, Adiponectin, Leptin and Ghrelin. Also at these point of time every patient underwent a psychosocial evaluation with life style questioners.

Safety:There were no complications with these modes of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Obese preadolescent children 6-11 year-old with BMI> 95th percentile for age and gender.
2. A signed informed consent will be taken from patients and their parents.
3. Agreement to a follow-up of one year.

Exclusion Criteria:

1. Cardiac problems (arrhythmia, Congestive heart disease)
2. Uncontrolled hypertension
3. Severe hepatic impairment (liver enzymes above 3 folds the upper normal values)
4. Renal failure
5. Genetic syndromes associated with obesity
6. Presence of untreated hypothyroidism
7. Participation in a clinical study during the last month

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160
Dates: Start 2004-04; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
BMI
BMI-SDS
BODY FAT PERCENTAGE
WAIST AND HIP CIRCUMFERENCES

SECONDARY OUTCOMES:
BLOOD METABOLIC PROFILE
BLOOD INFLAMATORY MARKERS
GHRELIN AND LEPTIN LEVELS
RESTING ENERGY EXPENDITURE
PSYCHOLOGICAL PARAMETERS

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, Prof, MD, Principal Investigator — Schneider Children Medical Center
Locations (2):
- Israel (2):
  - Soroka Medical Center, Beersheba
  - Schneider Children's Medical Center, Petah Tikva